CLINICAL TRIAL: NCT05944211
Title: A Randomized, Controlled Study on the Efficacy and Safety of Hetrombopag in the Treatment of Chemotherapy-induced Thrombocytopenia(CIT) in Patients With Acute Myeloid Leukemia
Brief Title: Hetrombopag for the Treatment of Chemotherapy-Induced Thrombocytopenia(CIT) in Patients With Acute Myeloid Leukemia
Acronym: H-CIT-AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-OBU-SH-CIT-II-001
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
Keywords: Chemotherapy-Induced Thrombocytopenia; Acute Myeloid Leukemia; Hetrombopag
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hetrombopag (Experimental): The study in a 1:1 randomization ratio (36 subjects to experimental group). The treatment group received Herteppa Ethanolamine tablets and platelet transfusion.
  Interventions: Drug: Hetrombopag Olamine
- Control (No Intervention): The study in a 1:1 randomization ratio (36 subjects to control group). The control group did not receive other platelet raising therapy except platelet transfusion.

INTERVENTIONS:
Drug: Hetrombopag Olamine — The subjects will initiate treatment with 7.5 mg hetrombopag once a day, starting orally 24 hours after the end of chemotherapy. Platelet counts is obtained weekly and dose adjustment should be done according to platelet counts once every two weeks, and maximum dose should not exceed 15 mg daily. Subjects whose platelet count <25×109/L for 2 weeks, the hetrombopag dose will be increased by 2.5mg. If subjects whose platelet count ≥100×109/L or who had received hetrombopag for 28 days, hetrombopag can be stopped. Hetrombopag Olamine is sponsored by Jiangsu Hengrui Pharmaceuticals Co., Ltd.
  Emergency treatment: When the platelet count was less than 20×109/L, platelet transfusion was given according to the evaluation of the investigator.
  Arms: Hetrombopag

SUMMARY:
Randomized, controlled, open study to evaluate the efficacy and safety of Hetrombopag in the treatment of chemotherapy-induced thrombocytopenia(CIT) in patients with acute myeloid leukemia

DETAILED DESCRIPTION:
This study is a prospective, single center, randomized, controlled and open clinical trial initiated by the researchers to evaluate the efficacy and safety of Hetrombopag in the treatment of thrombocytopenia caused by chemotherapy in acute myeloid leukemia. The study focuses on acute myeloid leukemia patients aged 18-70 who have completed induction chemotherapy and achieved complete remission, and have received ≤ 1 course of intensive therapy for consolidation. Patients were randomly divided into the treatment group and the control group through the random number table by 1:1. The treatment group received Hetrombopag and platelet transfusion, and the control group did not receive other platelet raising therapy except platelet transfusion. The study used the proportion of subjects with effective treatment during the randomized treatment period as the main efficacy indicator. 72 patients are planned to be enrolled, with treatment group and control group=1:1.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70;
* Participant with a histologically or cytologically confirmed acute myeloid leukemia in complete remission (PLT≥100×109/L) (except acute promyelocytic leukemia);
* Participant who have completed induction therapy and achieved complete remission, have received ≤1 course of intensive consolidation chemotherapy, and will continue to receive intensive consolidation or maintenance chemotherapy;
* Intensive chemotherapy after complete remission including: high-dose or medium-dose cytarabine chemotherapy (1-1.5g/m2 q12h×3 days), standard-dose chemotherapy (cytarabine combined with anthracycline/anthraquinones, HHT, pohyllotoxin, etc.);
* Participant whose Expected survival time ≥3 months, and who can receive at least 2 cycles of intensive chemotherapy;
* ECOG performance status <=2;
* Participants of childbearing age who agree to use reliable contraceptive methods;
* Patients signed the informed consent form and volunteered to participate in this study with good compliance;

Exclusion Criteria:

* Participant has any history of hematologic diseases other than chemotherapy-induced thrombocytopenia;
* Participant has a history of arterial or venous thrombosis within 6 months before screening (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism), or has clinical symptoms and medical history suggestive of thrombophilia;
* Participant has a history of severe cardiovascular disease within 6 months before screening, such as congestive heart failure (NYHA class III-IV), arrhythmia known to increase the risk of thromboembolism (atrial fibrillation), post-coronary stent implantation, angioplasty, or coronary artery bypass grafting;
* Known human immunodeficiency virus infection,or hepatitis C infection (if hepatitis B surface antigen is positive, or hepatitis B surface antigen is negative but hepatitis B core antibody is positive, HBV-DNA testing is required, if virus replication is suggested, the subject should be excluded);
* Abnormal liver function (TBL>3xULN; alanine aminotransferase [ALT] or aspartate aminotransferase [AST]>3xULN);
* Abnormal renal function with serum creatinine>1.5xULN or creatinine clearance ≤ 60 ml/min using Cockcroft-Gault estimated creatinine clearance;
* Pregnant or lactating women, or those planning to receive/give birth in the near 6 months;
* Participant participated in other clinical trials within 3 months before enrollment;
* Previous use of thrombopoietin receptor agonist (TPO-RA), recombinant human TPO, recombinant human interleukin-11(rhlL-11) within 1 month before screening;
* Received platelet transfusions within 3 days before enrollment;
* Patients with known or expected allergy or intolerance to the active ingredient or excipients of hetrombopag;
* Inability to understand the nature of the study or failure to obtain informed consent;
* The investigator considers that there are any other conditions that may prevent the subject from completing the study or present a significant risk to the subject;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Days that platelet count firstly rebound to 100×109/L | Randomization up to 28 days

SECONDARY OUTCOMES:
Days that platelet count firstly rebound to 50×109/L | Randomization up to 28 days
The median dose and duration of hetrombopag from starting treatment to platelet count ≥100×109/L | Randomization up to 28 days
The minimum platelet count at the chemotherapy cycle | Randomization up to 28 days
The lasting days of platelet count below 50×109/L at the chemotherapy cycle | Randomization up to 28 days
The lasting days of platelet count below 25×109/L at the chemotherapy cycle | Randomization up to 28 days
The number of platelet transfusions at the chemotherapy cycle | Randomization up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Han, MD.,Ph.D, Principal Investigator — RenJi Hospital; Yi Fang, MD.,Ph.D, Principal Investigator — RenJi Hospital